CLINICAL TRIAL: NCT04791930
Title: Evaluation of Vestibular Function in Patients With Chronic Suppurative Otitis Media: Safe Type
Brief Title: Evaluation of Vestibular Function in Patients With C.S.O.M: Safe Type
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed Abd Elhameed Ali, Principle Investigator, Assiut University
Other Study IDs: VNG&C.S.O.M
Record Dates: First submitted 2021-02-09; First posted 2021-03-10 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Vertigo Labyrinthine
Keywords: Chronic suppurative otitis media; safe type; vertigo; vestibular testing; vestibular function; VNG; Rotatory Chair
MeSH Terms: conditions — Vertigo

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

SUMMARY:
To evaluate the function of vestibular system in patients with chronic suppurative otitis media safe type.

DETAILED DESCRIPTION:
Chronic suppurative otitis media (CSOM) remains one of the most common chronic infectious diseases worldwide, affecting diverse racial and cultural groups both in developing and industrialized countries. It involves considerable morbidity and can cause extra- and intracranial complications .

CSOM in all its clinical presentations (acute, serous and chronic) develops with varying degrees of lesions in the inner ear, which showing a higher prevalence of disabling hearing loss, tinnitus and balance and vestibular alterations.

In recent years, authors have raised the hypothesis that the vestibular system could also be subject to inflammatory lesions secondary to CSOM. These hypotheses were supported by clinical studies, which disclosed a high prevalence of vestibular symptoms in patients with CSOM (40% -60%), in addition to changes in several vestibular function tests (caloric testing, rotary chair, vestibular evoked myogenic potentials, vHIT and posturography) .

Over the years, several studies have analyzed the potential clinical impact of CSOM on vestibular function (Monsanto et al, 2018). However, a recent systematic review showed that these studies are mostly have had several biases identified (selection, attrition, performance and detection) .

Also, there are a number of difficulties regarding changes in vestibular function secondary to CSOM, mainly because several vestibular function tests (caloric testing, vestibular evoked myogenic potentials) do not have validated results for patients with middle ear disorders inherent to CSOM (tympanic perforation, ossicular erosion, fibrosis or secretion in the middle ear, and conductive hearing loss), and therefore are not directly comparable to those of patients without middle ear diseases.

Furthermore, CSOM is more prevalent in the elderly, who have several other possible causal factors for vestibular symptoms, therefore, directly correlating CSOM with changes in vestibular function is a challenging task .

One of the vestibular function tests of that is not significantly influenced by CSOM is the video head impulse test, this test can objectively assess the function of each one of the semicircular canals alone, providing important information regarding changes in the vestibulo-ocular reflex (VOR), despite these advantages, the literature on the use of the video head impulse test in patients with COM is very scarce. Considering the role of the head impulse test in the diagnosis of VOR alterations, the identification of alterations in this test can help in the topographic characterization of vestibular alterations secondary to COM .

Evaluation of vestibular function in patients with safe type chronic suppurative otitis media provide many strategies aimed to prevent the sequelae and give idea about selection of adequate treatment and rehabilitation .

ELIGIBILITY:
Inclusion Criteria:

* Age: from 10 years to 45 years old.
* Sex: male or female.
* Safe type Chronic Suppurative Otitis Media.

Exclusion Criteria:

* Un safe type Chronic Suppurative Otitis Media.
* Noise exposure and heredofamilial hearing loss.
* Adhesive process or history of ear surgery.

Ages: 10 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: patients with chronic suppurative otitis media safe type.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-10-28 (Estimated); Primary Completion 2023-04-28 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Vestibular evaluation | Baseline
  The incidence and extent of vestibular dysfunction in patients with chronic suppurative otitis media: safe type

CONTACTS AND LOCATIONS:
Overall Officials: Enass sayed Mohamed, Professor, Principal Investigator — Assiut University
Locations (1):
- Assuit University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Monsanto RDC, Kasemodel ALP, Tomaz A, Elias TGA, Paparella MM, Penido NO. Evaluation of vestibular symptoms and postural balance control in patients with chronic otitis media. J Vestib Res. 2020;30(1):35-45. doi: 10.3233/VES-200691. PMID 32083607